CLINICAL TRIAL: NCT02707718
Title: Early Biomarkers of Sepsis Identification in the Emergency Department
Brief Title: Biomarkers for the Early Identification of Sepsis in the Emergency Department
Acronym: BIPS
Status: Completed | Type: Observational
Sponsor: Pitié-Salpêtrière Hospital (Other)
Collaborators: Institut Pasteur (Industry); Bio-Rad Laboratories (Industry)
Responsible Party: Principal Investigator, Hausfater Pierre, Principal investigator, Pitié-Salpêtrière Hospital
Other Study IDs: BIPS study
Record Dates: First submitted 2016-02-26; First posted 2016-03-14 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Sepsis
Keywords: sepsis; biomarker; prognostic; emergency department; diagnosis
MeSH Terms: conditions — Sepsis; Emergencies; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and sera
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood sampling — during the usual blood sampling performed in the ED in patients suspected of sepsis, two additional tubes will be sampled for a panel of biomarkers measurement

SUMMARY:
Monocentric prospective study on consecutive patients attending the emergency department and suspected to have sepsis. Blood sampling for the measurement of a panel of biomarkers of interest in sepsis.

DETAILED DESCRIPTION:
The management of patients admitted to the emergency department (ED) requires investigative biological parameters that help clinicians to make the right diagnosis.

Sepsis concerns patients with infection associated with a systemic inflammatory response. While this inflammatory profile is observed in many clinical situations in the ED, the challenge is to characterize in these patients suspected of sepsis those who have a real infection.

Currently, no individual biomarker of sepsis is sufficiently discriminant. The objective of this study is to measure in patients suspected of sepsis in the emergency department, a combination of biomarkers (covering several distinct pathophysiological pathways) that could provide high specificity and sensitivity for the diagnostic and prognostic. The originality of this study is that compared with patients admitted to intensive care units, patients investigated for suspected sepsis in the ED are seen earlier in their medical history and usually before any therapeutic intervention (intravenous fluids, antibiotics, catecholamines) interfering with several biomarkers of interest.

ELIGIBILITY:
Inclusion Criteria:

* patient attending the ED and suspected to have sepsis by the emergency physician after clinical exam

Exclusion Criteria:

* patient minor under 18-year
* pregnancy
* anticipated no follow-up possible (homeless...)
* Refusal to participate
* patient under curators, prisoner

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients attending the ED and suspected to have sepsis
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
sepsis diagnosis | 30-day after inclusion
  Among the patients included in the study with a sepsis suspicion, the primary outcome measure will be a final diagnosis of sepsis adjudicated on the medical file and 30-day follow-up, by an expert panel blind for the biomarkers studied

SECONDARY OUTCOMES:
severe outcome defined by: severe sepsis and/or septic shock and/or ICU admission and/or death in the 30-day follow-up | 30-day after inclusion
  Among the patients included in the study with a sepsis suspicion, a diagnosis of severe sepsis and/or septic shock will be adjudicated on the medical file and 30-day follow-up by an expert panel blind for the biomarkers studied. ICu admission and death will be recorded by the medical file and 30-day phone interview.

CONTACTS AND LOCATIONS:
Overall Officials: pierre Hausfater, Md PhD, Principal Investigator — ARCEAR
Locations (2):
- France (2):
  - Hôpital Pitié Salpêtrière, Paris
  - Institut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: No